CLINICAL TRIAL: NCT03948412
Title: Incision Management With Prevena After Renal Transplant (IMPART) Trial: Negative Pressure Wound Therapy Versus Standard Dressings for Incision Management After Renal Transplant: a Multicentre, Partially-blinded Randomised Controlled Trial
Brief Title: Negative Pressure Wound Therapy (PREVENA) Versus Standard Dressings for Incision Management After Renal Transplant
Acronym: IMPART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, David Herlihy, Vascular Surgery Registrar, Royal North Shore Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RNSH-VASC-2019-1
Record Dates: First submitted 2019-05-05; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Wound Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Closed Incision Negative Pressure Wound Therapy (Prevena) (Experimental): Patients are randomised intra-operatively to either Prevena or standard dressings as long as inclusion criteria are met, and no exclusion criteria met. This is left in-situ for 7 days, unless clinically indicated.
  Interventions: Device: Closed Incision Negative Pressure Wound Therapy (Prevena)
- Standard Dressings (Active Comparator): Patients are randomised intra-operatively to either Prevena or standard dressings as long as inclusion criteria are met, and no exclusion criteria met. Standard care wound dressings are applied for patients in this arm. These are changed as clinically appropriate whilst in hospital.
  Interventions: Other: Control - Standard Dressings

INTERVENTIONS:
Device: Closed Incision Negative Pressure Wound Therapy (Prevena) — Closed Incision Negative Pressure Wound Device (Prevena) applied to closed wound at completion of operation.
  Arms: Closed Incision Negative Pressure Wound Therapy (Prevena)
Other: Control - Standard Dressings — Standard wound dressings applied to closed wound at completion of operation.
  Arms: Standard Dressings

SUMMARY:
This study is a multicentre, partially-blinded randomised controlled trial, with site stratified block randomisation and partial blinding of outcome assessments. Patients undergoing a renal transplant will be allocated to one of two treatment arms, where either a Prevena device of appropriate size or standard dressing is applied to the closed incision. In the case that a patient requires bilateral incisions, both incisions will be allocated to the same treatment arm and counted as a single incision.

Primary:

The primary objective of this study is to determine if the Prevena Incision Management System reduces wound complications at the surgical site following renal transplant, when compared to standard dressings. Secondary: Secondary objectives of this study include identification of risk factors for wound complications at the surgical site, as well as re-operation, prolonged hospital stay, allograft survival, delayed graft function. This study will also assess pain, scar healing and quality of life in each treatment arm, and aim to complete a cost-benefit analysis of the Prevena device in renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

The participant:

1. is an adult ≥ 18 years old, regardless of comorbidities or BMI
2. is able to provide their own informed consent
3. will undergo open renal transplant surgery, including those who undergo dual renal transplant or simultaneous pancreas transplant.
4. will require a surgical incision(s) likely to be able to be covered completely by one or more Prevena Incision Management Systems.
5. is willing and able to return for the required follow up assessments.
6. if concurrently enrolled in a clinical trial it must not impact on patient health or the surgical incision site and the study must be documented

Exclusion Criteria:

The participant:

1. has a known allergy or hypersensitivity to silver, or drape materials that contain acrylic adhesives.
2. Is not suitable for closure of the surgical wound, and as such the wound must be left open or an open NPWT device is required.
3. Is not willing to comply with the study procedures.
4. Has an unforseen intraoperative event mandating additional management including a planned re-exploration.
5. Has obvious intraoperative contamination of the surgical site.
6. Has a wound with suspected ischaemia in the incision area, or inadequate haemostasis. 7. Requires drains that cannot be covered by the Prevena dressing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-05-10 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Wound Complications | 0-90 days
  Any wound infection, wound dehiscence, wound haematoma, wound collection or re-operation due to the above following renal transplantation.

SECONDARY OUTCOMES:
Length of hospital stay | 0-90 days
  Comparison of length of hospital stay between the two groups
Graft function (creatinine) | 0-90 days
  Comparison of markers of graft function (creatinine) between the two groups
Delayed graft function | 0-90 days
  Number of patients requiring ongoing dialysis in each group.
Pain score (numeric rating scale) | 0-90 days
  Comparison of patient reported post-operative wound pain scale between groups utilising a generic numeric rating scale (NRS) for pain.
  A numeric rating scale is a way a patient can report pain from 0-10, 0 being no pain, 10 being extreme pain. Minimum score is 0, maximum score is 10. It is better to have less pain, therefore 0 is the best score possible.
Scar quality (The Patient and Observer Scar Assessment Scale: POSAS) | 0-90 days
  Comparison of observer and patient reported scarring utilising the POSAS (The Patient and Observer Scar Assessment Scale: POSAS).
  The observer questions are listed below and are each scored from 1 to 10, 1 being normal skin, 10 being worst scar imaginable.
  1. Vascularity
  2. Pigmentation
  3. Thickness
  4. Relief
  5. Pliability
  6. Surface area
  7. Overall opinon of scar The patient scale questions are listed below and are each scored from 1 to 10, 1 being normal skin, 10 being the worst scar imaginable.
  1. Has the scar been painful the past few weeks? 2. Has the scar been itching the past few weeks? 3. Skin Colour 4. Skin stiffness 5. Skin Thickness 6. Scar irregularity 7. Overall opinion of scar The total score for patient and observer subscales is out of 70 each, for a combined total of 140 (both subscales added together). The minimum possible score is 14 and the maximum score is 140.
Quality of Life (EQ-5D-5L score) | 0-90days
  Comparison of quality of life scores reported by patients in each group using the EQ-5D-5L quality of life scale.
  The scale is split into 5 subscales;
  1. mobility
  2. self-care
  3. usual activities
  4. pain/discomfort
  5. anxiety/depression. Each subscale is ranked from 1 to 5, 1 being nil pain/quality of life disturbance, 5 being extreme pain/quality of life disturbance. The subscales are reported separately and are not combined.
  The patient also completes an overall health assessment from 0-100, 0 being the worst health imaginable, 100 being the best health imaginable. This is also reported and analysed separately.
Graft function (estimated glomerular filtration rate) | 0-90days
  Comparison of markers of graft function (creatinine) between the two groups
ASEPSIS wound score | 0-90days
  Wound scoring by a wound assessor.
  Scored:
  0-5 for serous discharge and erythema (each), 0 being nil, 5 being significant. 0-10 for purulent exudate and separation of deep tissues (each), 0 being nil, 10 being significant.
  Isolation of bacteria on wound swap, 0 for no bacterial, 10 for bacterial growth.
  Further scores of 10 (for antibiotic usage), 5 (for drainage of pus under local anaesthesia), 10 (for debridement under general anaesthesia) and 5 (for prolonged inpatient stay >14 days).
  All scores are added together for a total of 70, 0 being the minimum possible (best) score and 70 being the maximum possible (worst) score.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Puttaswamy, MBBS, Principal Investigator — Vascular Surgeon
Locations (1):
- Royal North Shore Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03948412/Prot_SAP_000.pdf